CLINICAL TRIAL: NCT01853215
Title: A Follow-Up Volunteer Study Evaluating Intraosseous Vascular Access Infusion in the Sternum Using the EZ-IO T.A.L.O.N.Intraosseous System.
Brief Title: Healthy Adult Volunteer Study of Intraosseous Infusion Using the Sternum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vidacare Corporation (Industry)
Responsible Party: Sponsor
Organization: Teleflex (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013-04
Record Dates: First submitted 2013-05-09; First posted 2013-05-14 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Intraosseous Vascular Access
Keywords: sternal intraosseous infusion study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sternal intraosseous vascular access (Experimental): Sternal intraosseous vascular access using T.A.L.O.N. Intraosseous System.
  Interventions: Device: T.A.L.O.N. Intraosseous System

INTERVENTIONS:
Device: T.A.L.O.N. Intraosseous System — intraosseous catheter for use in the sternum
  Other Names: EZ-IO TALON

SUMMARY:
This study is being done to evaluate intraosseous vascular access through the sternum.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the presence or absence of extravasation when using the T.A.L.O.N. Intraosseous System to establish sternal intraosseous infusion. This study will also evaluate the user preference feedback received from the device operators about the ease of use and level of satisfaction with the device. Lastly, this study will evaluate the infusion flow rates obtained when using intraosseous infusion in the sternum.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older;
* healthy adult subjects

Exclusion Criteria:

* Weight < 45kg;
* BMI greater or equal to 30 with absence of adequate landmarks or too much overlaying tissue, as determined by the PI;
* Imprisoned subjects;
* pregnant subjects;
* prior sternotomy;
* cognitively impaired subjects;
* fracture in target bone, or significant trauma to the site;
* excessive tissue and/or absence of adequate anatomical landmarks in target bone;
* infection in target area;
* IO insertion in past 48 hours or other significant orthopedic procedure in target bone;
* current use of anti-coagulants;
* previous adverse reaction to Lidocaine;
* current cardiac condition requiring pacemaker or anti-arrhythmic drugs
* previous adverse reaction to contrast dye
* Allergy to any food and drug
* History of impaired renal function
* History of impaired hepatic function
* History of cardiac disease
* History of pheochromocytoma

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry J Miller, MD, Principal Investigator — Vidacare Corporation
Locations (1):
- Bulverde-Spring Branch EMS, Spring Branch, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults aged 21 years and older were recruited to participate in the study.
Groups:
- Sternal Intraosseous Vascular Access: sternal intraosseous vascular access using T.A.L.O.N.
  T.A.L.O.N. Intraosseous System: intraosseous catheter for use in the sternum
Period: Overall Study
Arm/Group | Sternal Intraosseous Vascular Access
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sternal Intraosseous Vascular Access: sternal intraosseous vascular access using T.A.L.O.N. Sternal Manual Intraosseous Needle set
  T.A.L.O.N. Sternal Manual Intraosseous Needle set : intraosseous catheter for use in the sternum
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Occurrences of Extravasation During Infusion
Description: The number of participants with occurrence of extravasation during intraosseous infusion as evidenced by contrast injection into the intraosseous catheter, visualized under fluoroscopic imaging.
Time Frame: during 12 minutes of infusion
Measure: Number; unit: participants
Groups:
- Sternal Intraosseous Vascular Access: sternal intraosseous vascular access using T.A.L.O.N.
  T.A.L.O.N. Intraosseous System : intraosseous catheter for use in the sternum
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 24
participants | 2

2. Secondary Outcome: Stability of Locator
Description: Operator's perceived stability of the sternal locator once placed on the subject.
  1 to 5 scale was used with 1=Poor; 2=Fair; 3=Good; 4=Very good; 5=Excellent.
Time Frame: During insertion of the intraosseous needle set
Population: This outcome measure was not reported for one participant, thus only 23 participants were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Likert scale
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 23
Likert scale | 4.04 (1.15)

3. Secondary Outcome: Stability of Catheter Hub
Description: Ability to stabilize the catheter hub and rotate the stylet for removal. 1 to 5 scale was used with 1=Very difficult; 2-Difficult; 3=Neutral; 4=Easy; 5=Very easy.
Time Frame: During insertion of the intraosseous needle set
Measure: Mean (Standard Deviation); unit: Likert scale
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 24
Likert scale | 4.35 (0.8)

4. Secondary Outcome: Adhesion Strips
Description: Perceived effectiveness of the device adhesion strips after application. A 1- 5 scale was used with 1=Poor; 2=Fair; 3=Good; 4=Very good; 5=Excellent.
Time Frame: During insertion of the intraosseous needle set
Measure: Mean (Standard Deviation); unit: Likert scale
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 24
Likert scale | 3.83 (1.13)

5. Secondary Outcome: Gravity Flow Rates
Description: Measure the infusion flow rates attainable in the sternum when using intraosseous infusion of normal saline using a gravity infusion (no Pressure).
Time Frame: during the 12 minute infusion time frame
Population: One participant experienced a prior extravasation and therefore did not receive the gravity flowrate infusion. Only 23 participants were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 23
milliliters per hour | 1130.44 (691.79)

6. Secondary Outcome: 100 Millimeters of Mercury (mmHg) Infusion Flow Rates
Description: Measure the infusion flow rates attainable in the sternum when using intraosseous infusion of normal saline using a 100 mmHg infusion.
Time Frame: during the 12 minute infusion time frame
Population: One participant experienced a prior extravasation and therefore did not receive the 100 mmHG flowrate infusion. Only 23 participants were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 23
milliliters per hour | 3373.91 (1370.21)

7. Secondary Outcome: 200 Millimeters of Mercury (mmHg) Infusion Flow Rates
Description: Measure the infusion flow rates attainable in the sternum when using intraosseous infusion of normal saline using a 200 mmHg infusion.
Time Frame: during the 12 minute infusion time frame
Population: Two participants experienced a prior extravasation and therefore did not receive the 200 mmHg flowrate infusion. For one participant the 200 mmHg flowrate infusion was not performed. Therefore only 21 participants were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 21
milliliters per hour | 4619.05 (1785.39)

8. Secondary Outcome: 300 Millimeters of Mercury (mmHg) Infusion Flow Rates
Description: Measure the infusion flow rates attainable in the sternum when using intraosseous infusion of normal saline using a 300 mmHg infusion.
Time Frame: during the 12 minute infusion time frame
Population: Two subjects experienced a prior extravasation and therefore did not receive the 300 mmHg flowrate infusion. Thus only 22 subjects were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | Sternal Intraosseous Vascular Access
Number analyzed (Participants) | 22
milliliters per hour | 5327.27 (1724.39)

ADVERSE EVENTS:
Description: participants were monitored during study participation including a telephone follow-up call performed one day after the study procedure to assess for participant reported adverse events.
Arm/Group | Sternal Intraosseous Vascular Access
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes